CLINICAL TRIAL: NCT06724068
Title: The Correlation Between Diabetes, Insulin Resistance and Body Composition
Brief Title: Diabetes, Insulin Resistance and Body Composition
Status: Completed | Type: Observational
Sponsor: Xuan Song (Other)
Responsible Party: Sponsor-Investigator, Xuan Song, Principal Investigator, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: S1181
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Insulin Resistance, Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetes
  Interventions: Other: Diabetes，Insulin resistance，Control
- Insulin resistance
  Interventions: Other: Diabetes，Insulin resistance，Control
- Control
  Interventions: Other: Diabetes，Insulin resistance，Control

INTERVENTIONS:
Other: Diabetes，Insulin resistance，Control — This retrospective study uses medical records and diagnostic data from patients with type 2 diabetes and healthy controls obtained from Qianfoshan Hospital from2019 to 2022

SUMMARY:
The goal of this retrospective study is to learn about the correlation between diabetes, insulin resistance and body compositions.

The main question[s] it aims to answer are:

* [The difference of body composition between the individuals of insulin resistance and diabetes]
* [The effect of diabetes on body composition]

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older.
2. Diagnosed with type 2 diabetes mellitus according to recognized diagnostic criteria.
3. Availability of complete body composition data (e.g., DXA measurements).
4. Documented HbA1c levels and other glycemic control data.
5. Continuous medical records available during the study period

Exclusion Criteria:

1. Presence of other severe metabolic diseases, such as liver failure or kidney failure.
2. Use of medications affecting muscle mass (e.g., glucocorticoids) for more than three months.
3. History of malignancy or ongoing treatment for cancer.
4. Missing critical research data (e.g., diabetes duration or HbA1c levels).
5. History of surgeries causing significant body composition changes (e.g., bariatric surgery).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients aged 18 years and older who were diagnosed with type 2 diabetes mellitus. The population consists of individuals with documented medical records, including diabetes duration, glycemic control data (HbA1c levels), and body composition measurements such as muscle mass assessments. The study also includes a control group of non-diabetic individuals matched by age and sex to enable comparative analysis.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sarcopenia in Diabetic Patients | Retrospective analysis of data collected between2019 and 2022
  The proportion of diabetic patients diagnosed with sarcopenia, assessed based on measurements of muscle mass, muscle strength, and physical performance. Sarcopenia will be defined according to AWGS 2019 and EWGSOP2

CONTACTS AND LOCATIONS:
Overall Officials: Song Xuan, Doctor, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China